CLINICAL TRIAL: NCT04455815
Title: A Randomised Phase II Trial in Early COVID-19, Assessing Use of Camostat by Blocking SARS-CoV-2 Spike Protein-initiated Membrane Fusion.
Brief Title: A Trial Looking at the Use of Camostat in People Who Have Tested Positive for Coronavirus (COVID-19) (SPIKE-1)
Acronym: SPIKE-1
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Cancer Research UK (Other)
Collaborators: Latus Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CRUKD/20/002; 2020-002110-41 (EudraCT Number)
Record Dates: First submitted 2020-06-25; First posted 2020-07-02 (Actual); Results first posted 2023-12-11 (Actual); Last update posted 2023-12-11 (Actual); Status verified 2023-12

CONDITIONS: COVID-19 Infection
Keywords: COVID-19; Coronavirus Infections; Respiratory Tract Infections; Pneumonia, Viral; Virus Diseases; Camostat; Protease Inhibitors; Enzyme Inhibitors; Serine Proteinase Inhibitors
MeSH Terms: conditions — COVID-19; Coronavirus Infections; Respiratory Tract Infections; Pneumonia, Viral; Virus Diseases | interventions — camostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Camostat (Experimental): Patient to receive treatment with camostat tablets, 200mg four times daily (qds) for 14 days.
  Interventions: Drug: Camostat
- Control arm (No Intervention): Patient to receive best supportive care.

INTERVENTIONS:
Drug: Camostat — Patient to receive treatment with camostat tablets, 200mg four times daily (qds) for 14 days.
  Other Names: Camostat mesylate; Camostat mesilate
  Arms: Camostat

SUMMARY:
This is a phase II randomised, multicentre, prospective, open label clinical trial. The trial aims to recruit patients who test positive for COVID-19 who have mild symptoms and therefore can treat their symptoms in the community. Patients who test positive for COVID-19 at hospital may also be able to participate.

DETAILED DESCRIPTION:
Coronavirus-induced disease 2019 (COVID-19) caused by SARS-CoV-2 infection is a highly contagious disease with a high and unpredictable morbidity and mortality, for which there is currently no specific treatment. Progression from a mild fatigue, fever and cough, to severe respiratory failure requiring mechanical ventilation may occur 1 to 2 weeks into the disease. This provides a window of opportunity in which patients in the early phase of the disease could be treated with a disease-modifying agent, to halt disease progression, prevent hospital admissions with respiratory failure and prevent death.

Camostat is a serine protease inhibitor in clinical use in Japan since 1985 to treat patients with chronic pancreatitis (inflammation of the pancreas) and has an acceptable safety profile. Camostat has been shown to inhibit SARS-CoV-2 entry into epithelial cells in vitro. A trial of this repurposed drug for treatment of COVID-19 in humans is urgently required to assess its impact on disease progression to respiratory failure and whether it can reduce mortality.

This trial will recruit up to 100 patients. Patients will be randomised into a treatment arm (camostat tablets) or control arm (best supportive care). Community patients will be called daily at home for 14 days by the clinical trial team to collect symptoms and record the general well-being of the patient. For those patients recruited from hospital, visits will continue in hospital, where feasible, until discharge when home visits will be able to continue. The primary aim of this trial is to further assess the safety and toxicity profile of camostat to support integration into a Phase III trial. Secondary aims are to determine if camostat can reduce the clinical progression of COVID-19 and therefore the need for hospital admission and supplemental oxygen as well as include collection of patient reported health status, severity of symptoms and biological markers of the virus and confirm PK profile for the active metabolite of camostat. As the understanding of COVID-19 develops and improves, the inclusion criteria may be adapted to support the trial outcomes. Patients will be recruited through various settings which may include primary care 'COVID-19 hub' clinics, COVID-19 community-based testing centres, identification through other hospital departments, NHS digital, Test and Trace (or equivalent) or other clinical environments.

ELIGIBILITY:
Inclusion Criteria:

1. Patient willing and able to give informed consent
2. Adults, 18 years of age and above
3. Symptomatic COVID-19 infection
4. Evidence of current COVID-19 infection from a validated assay

Exclusion Criteria:

The patient may not enter the trial if ANY of the following apply:

1. Significant electrolyte disturbance (e.g. hyperkalaemia, potassium > site specific upper limit of normal)
2. Alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) and/or Alkaline Phosphatase (ALP) ≥ 2.5 x ULN
3. Any condition that, in the Investigator's opinion, would not make the patient a good candidate for the clinical trial or would prevent adequate compliance with trial therapy e.g. mild cognitive impairment (unable to follow instructions for self-assessment readings as assessed by the Investigator).
4. Patients on long term supplementary oxygen requirement (patients for whom hospital admission would not be considered e.g. care plan in the community is in place, are not excluded)
5. Known hypersensitivity to camostat
6. Platelet count <100 x 10^9/L
7. Co-enrolment with a Clinical Trial of an Investigational Medicinal Product (CTIMP) will not be permitted. Co-enrolment with a clinical investigation of a Medical Device or a non-interventional clinical study will be considered on a study-by-study basis and in discussion with the relevant Chief Investigators and Sponsors and industrial collaborators.
8. Co-enrolment involving non-interventional research (including questionnaire or tissue only studies) will be allowed provided this is not expected to affect the outcomes of both studies or place undue burden upon participants and their families.
9. Female patients who are able to become pregnant (or are already pregnant or lactating). However, those patients who are of child bearing potential and have a negative serum or urine pregnancy test before enrolment and agree to use two forms of contraception (one effective form plus a barrier method [oral, injected or implanted hormonal contraception and condom; intra-uterine device and condom; diaphragm with spermicidal gel and condom]) or agree to sexual abstinence*, effective from the first administration of camostat, throughout the trial and for 28 days afterwards are considered eligible.

   (*Abstinence is only considered to be an acceptable method of contraception when this is in line with the preferred and usual lifestyle of the subject. Periodic abstinence [e.g. calendar, ovulation, symptothermal, post-ovulation methods] and withdrawal are not acceptable methods of contraception.)
10. Male patients with partners of child-bearing potential (unless they agree to take measures not to father children by using a barrier method of contraception [condom plus spermicide] or to sexual abstinence* effective from the first administration of camostat, throughout the trial and for 28 days afterwards. Men with partners of child-bearing potential must also be willing to ensure that their partner uses an effective method of contraception for the same duration for example, hormonal contraception, intrauterine device, diaphragm with spermicidal gel or sexual abstinence). Men with pregnant or lactating partners must be advised to use barrier method contraception (for example, condom plus spermicidal gel) to prevent exposure of the foetus or neonate.

    (*Abstinence is only considered to be an acceptable method of contraception when this is in line with the preferred and usual lifestyle of the subject. Periodic abstinence [e.g. calendar, ovulation, symptothermal, post-ovulation methods] and withdrawal are not acceptable methods of contraception.)
11. Significant cardiovascular disease (as assessed via the participant's medical record and history) as defined by:

    1. History of congestive heart failure requiring therapy (New York Heart Association [NYHA] III or IV)
    2. History of unstable angina pectoris or myocardial infarction up to 6 months prior to trial entry
    3. Presence of severe valvular heart disease
    4. Presence of a ventricular arrhythmia requiring treatment

Known allergic reactions to components of camostat e.g., lactose intolerance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2020-09-23 (Actual); Primary Completion 2021-11-29 (Actual); Study Completion 2022-03-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Dhaliwal, Professor, Principal Investigator — The Royal Infirmary of Edinburgh
Locations (9):
- United Kingdom (9):
  - Chawton Park Surgery, Alton
  - The Royal Infirmary of Edinburgh, Edinburgh
  - Church Avenue Medical Group, Harrogate
  - John Radcliffe Hospital, Oxford
  - Preston Lantern Centre, Preston
  - Clarence Medical Centre, Rhyl
  - Trafalgar Medical Practice, Southsea
  - Velindre Hospital, Wales
  - Eynsham Medical Centre, Witney

IPD SHARING:
Plan to Share IPD: Yes
Individual de-identified patient data will be shared with researchers whose proposed use of the data is approved by a review committee of the Sponsor.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: All requests made within 5 years from end-of-trial will be considered; requests made subsequently will be considered where possible.
Access Criteria: When a request has been approved Cancer Research UK will provide access to the de-identified individual patient-level data and appropriate supporting information. A signed Data Sharing Agreement must be in place before accessing requested information. Requests should be submitted to drugdev@cancer.org.uk.

REFERENCES:
- [Background] Halford S, Wan S, Dragoni I, Silvester J, Nazarov B, Anthony D, Anthony S, Ladds E, Norrie J, Dhaliwal K; CDD SPIKE-1 Project Team. SPIKE-1: A Randomised Phase II/III trial in a community setting, assessing use of camostat in reducing the clinical progression of COVID-19 by blocking SARS-CoV-2 Spike protein-initiated membrane fusion. Trials. 2021 Aug 19;22(1):550. doi: 10.1186/s13063-021-05461-9. PMID 34412682
- See also: A lay summary of the trial on the Health Research Authority website — https://www.hra.nhs.uk/planning-and-improving-research/application-summaries/research-summaries/spike-1-covid-19/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Trial participants were enrolled at four trial sites between 23 September 2020 and 23 June 2021.
Period: Randomisation Phase
Arm/Group | Camostat | Control Arm
Started | 16 | 18
Completed | 15 | 18
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0
Period: Treatment Phase
Arm/Group | Camostat | Control Arm
Started | 15 | 18
Completed | 13 | 16
Not Completed | 2 | 2
Not completed — Adverse Event | 0 | 1
Not completed — Hospital admission and treatment stopped in hospital | 1 | 0
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Camostat | Control Arm | Total
Number analyzed (Participants) | 16 | 18 | 34
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 14 | 15 | 29
  >=65 years | 2 | 3 | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 10 | 19
  Male | 7 | 8 | 15
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian / Asian British- Indian | 0 | 1 | 1
  Asian / Asian British- Pakistani | 0 | 1 | 1
  White- English / Welsh / Scottish / Northern Irish / British | 15 | 15 | 30
  Any other White background | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United Kingdom | 16 | 18 | 34

OUTCOME MEASURES:

1. Primary Outcome: Number of Camostat Related AEs and SAEs.
Description: Number of AEs and SAEs assessed as related to camostat by the Investigator.
Time Frame: Days 1 - 28
Population: All enrolled patients who received at least one dose of camostat. As only participants in the Camostat Arm received camostat, this outcome measure is reported in the Camostat Arm only.
Measure: Number; unit: Adverse Events
Arm/Group | Camostat
Number analyzed (Participants) | 16
Adverse Events
  Total AEs related to Camostat | 11
  Total SAEs related to Camostat | 0

2. Primary Outcome: Number of AEs by Severity Grade
Description: Number of AEs by Severity Grade (mild, moderate, severe)
Time Frame: Days 1 - 28
Population: All enrolled patients who received at least one dose of camostat (or complete Day 1 of the control arm).
Measure: Number; unit: Adverse Events
Arm/Group | Camostat | Control Arm
Number analyzed (Participants) | 16 | 18
Adverse Events
  Total Mild AEs | 25 | 25
  Total Moderate AEs | 10 | 5
  Total Severe AEs | 2 | 2
  Total Mild AEs related to Camostat | 5 | NA — Patients in the control arm received best supportive care. These patients did not receive camostat and so a relatedness assessment to camostat is not applicable.
  Total Moderate AEs related to Camostat | 6 | NA — Patients in the control arm received best supportive care. These patients did not receive camostat and so a relatedness assessment to camostat is not applicable.
  Total Severe AEs related to Camostat | 0 | NA — Patients in the control arm received best supportive care. These patients did not receive camostat and so a relatedness assessment to camostat is not applicable.

3. Secondary Outcome: PK Parameter Maximum Concentration (Cmax) of 4-(4-Guanidinobenzoyloxy)Phenylacetic Acid (GBPA).
Description: Maximum concentration (Cmax) of GBPA as assessed by population estimates from population PK analysis.
Time Frame: Days 7 and 14
Population: Analysis was not completed because no samples were collected for this analysis.
Arm/Group | Camostat | Control Arm
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: PK Parameter Time to Maximum Concentration (Tmax) of GBPA
Description: Time to maximum concentration (Tmax) of GBPA, as assessed by population estimates from population PK analysis.
Time Frame: Days 7 and 14
Population: Analysis was not completed because no samples were collected for this analysis
Arm/Group | Camostat | Control Arm
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: PK Parameter Area Under the Curve (AUC) of GBPA
Description: Area under the curve (AUC) of GBPA, as assessed by population estimates from population PK analysis.
Time Frame: Days 7 and 14
Population: Analysis was not completed because no samples were collected for this analysis
Arm/Group | Camostat | Control Arm
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: PK Parameter to Confirm Half-life (T1/2) of GBPA
Description: Half-life (T1/2) of GBPA as assessed by population estimates from population PK analysis
Time Frame: Days 1 - 28
Population: Analysis was not completed because no samples were collected for this analysis
Arm/Group | Camostat | Control Arm
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Number of Community Patients Admitted to Hospital Due to COVID-19
Description: Number of patients who were recruited in community healthcare settings who were subsequently admitted to hospital due to COVID-19.
Time Frame: Days 1 - 28
Population: Treatment arm patients who received camostat for a minimum of five days, and control arm patients who completed up to Day 14 or came off trial at an earlier timepoint due to an endpoint (e.g. hospitalisation).
Measure: Count of Participants; unit: Participants
Arm/Group | Camostat | Control Arm
Number analyzed (Participants) | 14 | 18
Participants | 2 | 3

8. Secondary Outcome: Number of Oxygen Free Days
Description: Number of days from Day 1 that each patient did not supplementary oxygen (median and range).
Time Frame: Days 1 - 28
Population: as for outcome 7
Measure: Median (Full Range); unit: Days
Arm/Group | Camostat | Control Arm
Number analyzed (Participants) | 14 | 18
Days | 28 [4 to 28] | 28 [0 to 28]

9. Secondary Outcome: Number of Ventilator - Free Days
Description: Number of days from Day 1 that each patient did not require ventilation (median and range).
Time Frame: Days 1 - 28
Population: as for outcome 7
Measure: Median (Full Range); unit: Days
Arm/Group | Camostat | Control Arm
Number analyzed (Participants) | 14 | 18
Days | 28 [28 to 28] | 28 [28 to 28]

10. Secondary Outcome: Time to Worst Point on the Scale or Deterioration of Two Points or More (From Randomisation) on 9 Point Category Ordinal Scale Ranging From '0 - Uninfected, no Clinical or Virological Evidence of Infection' to '8 - Death'
Description: Median time and range to worst point on the scale or deterioration of two points or more (from randomisation) on 9 point category ordinal scale. The scale was described in the protocol as follows: '0 - Uninfected, no clinical or virological evidence of infection, 1 - Ambulatory, no limitation of activities, 2 - Ambulatory, limitation of activities, 3 - Hospitalised - mild disease, no oxygen therapy, 4 - Hospitalised - mild disease, oxygen by mask or nasal prongs, 5 - Hospitalised - severe disease, non-invasive, ventilation or high-flow oxygen, 6 - Hospitalised - severe disease, intubation and mechanical ventilation, 7 - Hospitalised - severe disease, ventilation and additional organ support - vasopressors, renal replacement therapy (RRT), extracorporeal membrane oxygenation (ECMO), 8 - Death'
Time Frame: Days 1 - 28
Population: as for outcome 7
Measure: Median (Full Range); unit: Days
Arm/Group | Camostat | Control Arm
Number analyzed (Participants) | 14 | 18
Days | 0 [0 to 7] | 0 [0 to 7]

ADVERSE EVENTS:
Time Frame: Safety data was collected from the time of informed consent until 28 days from Day 1.Patients who were hospitalised were followed up for up to 28 days after they were discharged.
Description: AE terms from vocabulary, MedDRA V24.0.
Arm/Group | Camostat | Control Arm
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/18
Serious Adverse Events (participants affected / at risk) | 4/16 | 1/18
Other Adverse Events (participants affected / at risk) | 14/16 | 13/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Camostat (N=16) | Control Arm (N=18)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Oxygen saturation decreased (Investigations) | 3 (3) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Camostat (N=16) | Control Arm (N=18)
Alanine aminotransferase increased (Investigations) | 1 (1) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 1 (1) | 1 (1)
Chest discomfort (General disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Fibrin D dimer increased (Investigations) | 5 (5) | 7 (7)
Gamma-glutamyltransferase increased (Investigations) | 2 (2) | 4 (4)
Haemoglobin decreased (Investigations) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 2 (2) | 3 (3)
Lower respiratory tract infection bacterial (Infections and infestations) | 0 (0) | 1 (1)
Mouth ulceration (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 1 (1) | 0 (0)
Platelet count increased (Investigations) | 1 (1) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Swollen tongue (Gastrointestinal disorders) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Troponin increased (Investigations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Viral rash (Infections and infestations) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-09-20): https://cdn.clinicaltrials.gov/large-docs/15/NCT04455815/Prot_000.pdf
  • Statistical Analysis Plan (2022-03-03): https://cdn.clinicaltrials.gov/large-docs/15/NCT04455815/SAP_001.pdf